CLINICAL TRIAL: NCT06303115
Title: A Multi Site, Open Label, Parallel Group Study to Assess Changes in Tobacco Related Biomarkers of Exposure Following Switching From Smoking of Combustible Cigarettes to Exclusive Use of Nicotine Pouches in Adult Smokers
Brief Title: CSD231005 Nicotine Pouch Biomarkers of Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSD231005 BoE
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-03

CONDITIONS: Tobacco Use; Smoking
MeSH Terms: conditions — Tobacco Use; Smoking | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Nicotine Pouch P1312914, 4 mg nicotine (Active Comparator): Subjects will be switched to exclusive use of their assigned pouch flavor and strength.
  Interventions: Other: Nicotine Pouch P1312914, 4 mg nicotine
- Nicotine Pouch P1312915, 8 mg nicotine (Active Comparator): Subjects will be switched to exclusive use of their assigned pouch flavor and strength.
  Interventions: Other: Nicotine Pouch P1312915, 8 mg nicotine
- Nicotine Pouch P1013215, 8 mg nicotine (Active Comparator): Subjects will be switched to exclusive use of their assigned pouch flavor and strength.
  Interventions: Other: Nicotine Pouch P1013215, 8 mg nicotine
- Nicotine Pouch P1013218, 10 mg nicotine (Active Comparator): Subjects will be switched to exclusive use of their assigned pouch flavor and strength.
  Interventions: Other: Nicotine Pouch P1013218, 10 mg nicotine
- Nicotine Pouch P1012919, 12 mg nicotine (Active Comparator): Subjects will be switched to exclusive use of their assigned pouch flavor and strength.
  Interventions: Other: Nicotine Pouch P1012919, 12 mg nicotine
- Smoking Abstinence (Other): Subjects will not use any tobacco or nicotine containing products.
  Interventions: Other: Smoking Abstinence
- Continued UB cigarette smoking (Other): Subjects will continue use of their Usual Brand Cigarettes.
  Interventions: Other: Continued UB cigarette smoking

INTERVENTIONS:
Other: Nicotine Pouch P1312914, 4 mg nicotine — P1312914 pouch product
  Arms: Nicotine Pouch P1312914, 4 mg nicotine
Other: Nicotine Pouch P1312915, 8 mg nicotine — P1312915 pouch product
  Arms: Nicotine Pouch P1312915, 8 mg nicotine
Other: Nicotine Pouch P1013215, 8 mg nicotine — P1013215 pouch product
  Arms: Nicotine Pouch P1013215, 8 mg nicotine
Other: Nicotine Pouch P1013218, 10 mg nicotine — P1013218 pouch product
  Arms: Nicotine Pouch P1013218, 10 mg nicotine
Other: Nicotine Pouch P1012919, 12 mg nicotine — P1012919 pouch product
  Arms: Nicotine Pouch P1012919, 12 mg nicotine
Other: Smoking Abstinence — No tobacco/nicotine
  Arms: Smoking Abstinence
Other: Continued UB cigarette smoking — Usual Brand Cigarette
  Arms: Continued UB cigarette smoking

SUMMARY:
This will be a multi center open label, randomized, controlled, switching parallel-group study designed to assess changes in select biomarkers of exposure (BoE) in generally healthy smokers following a 5 day in-clinic switch to use of nicotine Pouch investigational products (IPs) compared to continued usual brand (UB) cigarette smoking or smoking abstinence.

ELIGIBILITY:
Inclusion Criteria:

Able to read, understand, and be willing to sign an Informed Consent Form (ICF) and complete questionnaires written in English.

Generally healthy males or females, 21 to 60 years of age, inclusive, at the time of consent.

Smokes combustible, filtered, nonmenthol or menthol cigarettes, 83 mm to 100 mm in length.

Smokes an average of at least 10 cigarettes per day (CPD) and inhales the smoke for at least six months prior to Screening. Brief periods of abstinence due to illness, a quit attempt (prior to 30 days of Screening), or clinical study participation (prior to 30 days of Screening) will be allowed at the discretion of the PI.

Self-reports that cigarettes are their primary tobacco- or nicotine-containing product use within 30 days of Screening. (Note: occasional use of other tobacco- or nicotine-containing products may be acceptable in consultation with the Sponsor);

Agrees to use assigned IP throughout the study period.

Expired breath carbon monoxide (ECO) level ≥ 10 ppm and ≤ 100 ppm at Screening and at CheckIn on Day 2.

Positive urine cotinine test at Screening.

Response at Screening to the Fagerström Test for Nicotine Dependence (FTND) question 1 ("How soon after you wake up do you smoke your first cigarette?") is either "Within 5 minutes" or "630 minutes." (Heatherton, Kozlowski, Frecker, & Fagerstrom, 1991).

Willing to switch from current UB cigarette to either nicotine Pouch IP, or abstain from smoking, for approximately 5 days during in-clinic confinement;

Females must be willing to use a form of contraception acceptable to the PI from the time of signing the informed consent until the End of Study (EOS).

Examples of acceptable means of birth control are, but not limited to:

1. Surgical sterilization (hysterectomy, bilateral tubal ligation/occlusion, bilateral oophorectomy, bilateral salpingectomy);
2. Established use of oral, implantable, injectable or transdermal methods of contraception associated with inhibition of ovulation (see Section 6.10 regarding the use of hormonal methods of contraception in females aged ≥ 35);
3. Physical barrier method (e.g., condom, diaphragm/sponge/cervical cap) with spermicide;
4. Non-hormone releasing intrauterine devices (IUD) or hormone-releasing IUDs (e.g., Mirena or Kyleena) (see Section 6.10 regarding the use of hormonal methods of contraception in females aged ≥ 35);
5. Vasectomized partner;
6. Abstinence from heterosexual intercourse (as a lifestyle choice, not just for the purpose of study participation); and
7. Post-menopausal and not on hormone replacement therapy.

Males must be willing to use a barrier method of contraception (e.g., a condom with spermicide) or to refrain from donating sperm from the time of signing the informed consent until the EOS, unless they had undergone a vasectomy or were abstinent from heterosexual intercourse, or their female partner was not able to bear children.

Willing to refrain from consuming cruciferous vegetables and grilled, smoked, fried or barbequed food, and to avoid being in the presence of the cooking of these foods. Subjects should also be willing to refrain from consuming cured sandwich meats, bacon, salami, and sausages 48 hours prior to CheckIn on Day 2.

Agrees to inclinic confinement of 8 days (7 nights).

Exclusion Criteria:

The presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the subject unsuitable to participate in this clinical study.

History, presence of, or clinical laboratory test results indicating diabetes. Fasting plasma glucose > 126 mg/dL (7 mmol/L) is exclusionary. One recheck may be performed for fasting plasma glucose values > 126 mg/dL but < 200 mg/dL.

Scheduled treatment for asthma currently or within the past 12 consecutive months prior to Screening. As needed treatment, such as inhalers, may be included at the PI's discretion, pending approval from the Medical Monitor.

Use of any medications that interfere with the cyclooxygenase pathway (e.g., antiinflammatoryanti-inflammatory drugs such as aspirin and ibuprofen) 14 days prior to CheckIn on Day 2.

Use of medications or substances (other than nicotine) known to be strong inducers or inhibitors of cytochrome P450 (CYP) enzymes within 14 days or 5 halflives of the medication or substances (whichever is longer) prior to CheckIn on Day 2.

History or presence of bleeding or clotting disorders.

Any history of cancer, except for primary cancers of the skin, such as localized basal cell/squamous cell carcinoma, that have been surgically and/or cryogenically removed.

Systolic blood pressure (BP) of > 160 mmHg or a diastolic BP of > 95 mmHg, measured after being seated for 5 minutes at Screening and CheckIn on Day 2.

Body Mass Index (BMI) < 18.0 or >40.0 kg/m2 (weight of ≤ 110 pounds) at Screening.

Hemoglobin level < 12.5 g/dL for females or <13.0 g/dL for males at Screening.

Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.

A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at Screening or CheckIn on Day 2.

Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBbsAg), or hepatitis C virus (HCV).

Use of any medication or substance that aids in smoking cessation, including but not limited to any NRT (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to signing of the ICF.

Postpones a decision to quit using tobacco or nicotinecontaining products to participate in this study or has made a previous quit attempt within (≤) 30 days prior to the signing of the ICF.

Any daily use of aspirin (≥ 325 mg/day) or anticoagulants (e.g., Clopidogrel [Plavix®], Warfarin [Coumadin®, Jantoven®]).

Individuals ≥ 35 years of age currently using systemic, estrogencontaining contraception or hormone replacement therapy.

Whole blood donation within 8 weeks (≤ 56 days) prior to the signing of the ICF.

NOTE: Subjects will be advised against scheduling a whole blood donation for at least 7 days following study completion.

Plasma donation within (≤) 7 days prior to the ICF. NOTE: Subjects will be advised against scheduling a plasma donation for at least 7 days following study completion.

Employed by a tobacco or nicotine company, the study site, or handles tobacco or nicotinecontaining products as part of their job.

Participation in another clinical trial within (≤) 30 days prior to the signing of the ICF. The 30day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the ICF in the current study.

Drinks more than 21 servings of alcoholic beverages per week.

Has a positive alcohol result at Screening or CheckIn on Day 2.

Determined by the PI to be inappropriate for this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2024-08-22 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
4(methylnitrosamino)1(3pyridyl)1butanol [NNAL] + glucuronides [Total NNAL] | 24 hour

SECONDARY OUTCOMES:
4Aminobiphenyl [4ABP] | 24 hour
1Aminonaphthalene [1AN] | 24 hour
2Aminonaphthalene [2AN] | 24 hour
2Cyanoethyl mercapturic acid [CEMA] | 24 hour
3Hydroxypropyl mercapturic acid [3HPMA] | 24 hour
3Hydroxy1methylpropylmercapturic acid [HMPMA] | 24 hour
3hydroxybenzo[a]pyrene [3-OH-B[a]P] | 24 hour
1hydroxypyrene [1OHP] | 24 hour
Monohydroxybutyl mercapturic acid [MHBMA] | 24 hour
Nnitrosonornicotine [NNN] + glucuronides [Total NNN] | 24 hour
SPhenyl mercapturic acid [SPMA] | 24 hour
Total nicotine equivalents (molar sum of nicotine, cotinine, 3hydroxycotinine and their glucuronides) [TNneq] | 24 hour
Carboxyhemoglobin [COHb] | 12 hour
Nnitrosonornicotine [NNN] + glucuronides [Total NNN] | 12 hour

CONTACTS AND LOCATIONS:
Overall Officials: Brian Keyser, PhD, Principal Investigator — Reynolds American
Locations (5):
- United States (5):
  - Pillar Bentonville, Bentonville, Arkansas
  - AMR Lexington, Lexington, Kentucky
  - QPS Missouri, Springfield, Missouri
  - AMR Knoxville, Knoxville, Tennessee
  - Pillar Richardson, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No